CLINICAL TRIAL: NCT01130532
Title: Tadalafil Once Daily Following As-Needed Phosphodiesterase Type 5 Inhibitor Treatment, an Assessment of Return to Normal Erectile Function
Brief Title: A Study in Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13461; H6D-US-LVIP (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2012-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; ED; Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2.5 milligram (mg) titrated to 5 mg Tadalafil (Active Comparator): 2.5 mg for 4 weeks, followed by 5 mg for 8 weeks with option to continue treatment at 5 mg for an additional 4 weeks
  Interventions: Drug: Tadalafil
- 5 mg Tadalafil (Active Comparator): 5.0 mg for 12 weeks with option to continue treatment for additional 4 weeks
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Administer orally
  Other Names: Cialis; LY450190
  Arms: 2.5 milligram (mg) titrated to 5 mg Tadalafil; 5 mg Tadalafil
Drug: Placebo — Administer orally
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate if treatment with tadalafil once daily will allow men to return to normal erectile function in those who did not have normal erectile function following as-needed (PRN) Phosphodiesterase Type 5 (PDE5) Inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least a 3-month history of erectile dysfunction (ED).
* Are able to read, understand and provide signed informed consent.
* Have an International Index of Erectile Function-Erectile Function (IIEF-EF) domain score that is greater than or equal to 17 and less than 26 at screening.
* Have been taking a maximum dose of sildenafil citrate (100 milligram [mg]), vardenafil (20 mg), or tadalafil (20 mg) on as needed basis for at least one month prior to screening.
* Anticipate having the same female sexual partner during the study who is willing to participate in the required number of sexual intercourse attempts and complete study measures during the study.
* Agree to make at least four sexual intercourse attempts during both the 4-week as needed run-in period and the 4-week non-drug run-in period.
* Agree not to use any other erectile dysfunction (ED) treatment, including herbal therapy during the 4-week non-drug, run-in, the double-blind treatment period, the open label period and for 96 hours after the end of the study.

Partner Inclusion Criteria:

* Are female and at least 18 years of age at screening.
* Anticipate having the same male study subject as her sexual partner during the study.
* Able to read, understand and provide signed informed consent.
* Agree to make the required number of sexual intercourse attempts with the male sexual study partner during the study.
* Willing to participate in recording responses to the treatment satisfaction scale.

Exclusion Criteria:

* Have an IIEF-EF domain score of greater than or equal to 26 at screening.
* Prior ineffective treatment with (or nonresponder to) any PDE5 Inhibitor
* Have previously used or are currently using any PDE5 inhibitor once daily.
* Present with ED caused by other primary disorders or ED caused by untreated/inadequately treated endocrine disease.
* Partner unwilling to complete all study requirements.
* History of radical prostatectomy or other pelvic surgery or penile implant, or a clinically significant penile deformity, in the opinion of the investigator
* Exhibit evidence of clinically significant renal insufficiency or hepatobiliary disease, or significant cardiac history as determined by the investigator
* Currently receive treatment with nitrates, cancer chemotherapy, or antiandrogens
* Have previously completed or withdrawn from this study or any other study investigating tadalafil for once-daily use.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (34):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newport Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tarzana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nampa, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poughkeepsie, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyndhurst, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bala-Cynwyd, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anderson, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mt. Pleasant, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Langley, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North York, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Kim E, Seftel A, Goldfischer E, Baygani S, Burns P. Comparative efficacy of tadalafil once daily in men with erectile dysfunction who demonstrated previous partial responses to as-needed sildenafil, tadalafil, or vardenafil. Curr Med Res Opin. 2015 Feb;31(2):379-89. doi: 10.1185/03007995.2014.989317. Epub 2014 Dec 2. PMID 25455432
- [Derived] Kim ED, Seftel AD, Goldfischer ER, Ni X, Burns PR. A return to normal erectile function with tadalafil once daily after an incomplete response to as-needed PDE5 inhibitor therapy. J Sex Med. 2014 Mar;11(3):820-30. doi: 10.1111/jsm.12253. Epub 2013 Jul 10. PMID 23841532

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 4 periods. Period I was a 4-week, as needed, run-in period. Period II was a 4-week, non-drug, wash-out period. Period III was a 12-week (Weeks 0-12), double-blind treatment. Period IV was a 4-week (Weeks 13-16), open-label treatment extension. Only participants completing Period III were eligible to continue into Period IV.
Groups:
- 2.5 mg Titrated to 5 mg Tadalafil: 2.5 milligram (mg) Tadalafil for 4 weeks, followed by 5 mg Tadalafil for 8 weeks during double-blind treatment period.
- 5 mg Tadalafil: 5.0 mg Tadalafil for 12 weeks during double-blind treatment period.
- Placebo: Placebo for 12 weeks during double-blind treatment period.
- 5 mg Tadalafil Open-Label Extension: 5 mg Tadalafil for 4 weeks during open-label treatment extension period.
Period: Period III (Weeks 0-12)
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil | 5 mg Tadalafil | Placebo | 5 mg Tadalafil Open-Label Extension
Started | 207 | 207 | 209 | 0
Received at Least 1 Dose of Study Drug | 205 | 205 | 207 | 0
Completed | 186 | 189 | 190 | 0
Not Completed | 21 | 18 | 19 | 0
Not completed — Adverse Event | 3 | 3 | 2 | 0
Not completed — Entry Criteria Not Met | 4 | 2 | 4 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 3 | 4 | 2 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 6 | 0
Period: Period IV (Weeks 13-16)
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil | 5 mg Tadalafil | Placebo | 5 mg Tadalafil Open-Label Extension
Started | 0 | 0 | 0 | 562 (Three participants who completed Period III chose not to continue into Period IV.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 546
Completed | 0 | 0 | 0 | 552
Not Completed | 0 | 0 | 0 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil | 5 mg Tadalafil | Placebo | Total
Number analyzed (Participants) | 207 | 207 | 209 | 623
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.68) | 58.1 (10.36) | 57.6 (10.17) | 57.6 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 207 | 207 | 209 | 623
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 9 | 27
  Not Hispanic or Latino | 199 | 197 | 200 | 596
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 2 | 2 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 29 | 24 | 35 | 88
  White | 173 | 177 | 167 | 517
  More than one race | 3 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 199 | 195 | 191 | 585
  Canada | 8 | 11 | 18 | 37
  Puerto Rico | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Having an International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score Greater Than or Equal to 26 Through 12-Week Endpoint (Double-Blind Treatment Period)
Description: Self-reported erectile function over the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Data presented are the percentage of participants who return to normal erectile function (IIEF-EF domain score ≥26) at end of double-blind treatment period (Period III).
Time Frame: Baseline through 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline IIEF-EF measurement, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Number; unit: percentage of participants
Groups:
- 2.5 mg Titrated to 5 mg Tadalafil (Period III): 2.5 milligram (mg) Tadalafil for 4 weeks, followed by 5 mg Tadalafil for 8 weeks during double-blind treatment period (Period III).
- 5 mg Tadalafil (Period III): 5.0 mg Tadalafil for 12 weeks during double-blind treatment period (Period III).
- Placebo (Period III): Placebo for 12 weeks during double-blind treatment period (Period III).
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 194 | 197 | 199
percentage of participants | 38.7 | 39.6 | 12.1
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, Fisher Exact

2. Secondary Outcome: Change From Baseline to 12-Week Endpoint in the International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score
Description: Self-reported erectile function over the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 194 | 197 | 199
units on a scale | 7.9 (0.49) | 8.1 (0.49) | 1.8 (0.49)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 6.1, Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 6.2, Standard Error of Mean 0.68

3. Secondary Outcome: Change From Baseline to 12-Week Endpoint in the International Index of Erectile Function - Intercourse Satisfaction (IIEF-IS) Domain Score
Description: Self-reported intercourse satisfaction over the past 4 weeks. IIEF-IS is the sum of Questions 6, 7 and 8 of the IIEF. Scores range from 0 (low/no satisfaction) to 5 (high satisfaction) for each question, with the total possible score for the 3 questions of 0 to 15. Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline IIEF-IS measurement, excluding those with International Index of Erectile Function - Erectile Function (IIEF-EF) domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 194 | 197 | 198
units on a scale | 2.8 (0.21) | 2.6 (0.21) | 0.6 (0.21)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 2.1, Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 2.0, Standard Error of Mean 0.29

4. Secondary Outcome: Change From Baseline to 12-Week Endpoint in the International Index of Erectile Function - Overall Satisfaction (IIEF-OS) Domain Score
Description: Self-reported overall satisfaction over the past 4 weeks. IIEF-OS is the sum of Questions 13 and 14; each question scored as 1 (low/no satisfaction) through 5 (high satisfaction) with total subscore for the 2 questions of 2 to 10. Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline IIEF-OS measurement, excluding those with International Index of Erectile Function - Erectile Function (IIEF-EF) domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 194 | 197 | 199
units on a scale | 2.4 (0.16) | 2.4 (0.16) | 0.6 (0.16)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 1.7, Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 1.7, Standard Error of Mean 0.22

5. Secondary Outcome: Change From Baseline to 12-Week in Percentage of "Yes" Responses to Sexual Encounter Profile (SEP) Questions 1-5
Description: Assessed was the mean change from baseline in the percentage of Yes responses to the SEP diary Questions 1-5. Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline SEP Questions assessment, excluding those with International Index of Erectile Function - Erectile Function (IIEF-EF) domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: percentage of "yes" responses
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 193 | 195 | 196
percentage of "yes" responses
  Question 1: Able to Achieve Erection | 12.2 (1.63) | 11.4 (1.62) | 1.8 (1.62)
  Question 2: Able to Insert | 26.2 (2.25) | 26.1 (2.23) | 6.9 (2.23)
  Question 3: Successful Intercourse | 37.3 (2.52) | 39.4 (2.50) | 12.6 (2.51)
  Question 4: Satisfied with Hardness | 44.2 (2.73) | 42.8 (2.70) | 11.5 (2.71)
  Question 5: Overall Satisfaction with Experience | 43.6 (2.70) | 41.2 (2.68) | 10.6 (2.68)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Question 1. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 10.4, Standard Error of Mean 2.28
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = 9.6, Standard Error of Mean 2.26
Statistical Analysis 3: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Question 2. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 19.3, Standard Error of Mean 3.14
Statistical Analysis 4: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 3]; LS Mean Difference = 19.3, Standard Error of Mean 3.12
Statistical Analysis 5: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Question 3. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 24.7, Standard Error of Mean 3.53
Statistical Analysis 6: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 5]; LS Mean Difference = 26.8, Standard Error of Mean 3.50
Statistical Analysis 7: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Question 4. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 32.7, Standard Error of Mean 3.82
Statistical Analysis 8: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 7]; LS Mean Difference = 31.3, Standard Error of Mean 3.79
Statistical Analysis 9: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Question 5. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 33.0, Standard Error of Mean 3.78
Statistical Analysis 10: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 5, analysis 9]; LS Mean Difference = 30.5, Standard Error of Mean 3.75

6. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Treatment Satisfaction Scale (TSS) - Patient
Description: The TSS measured participant satisfaction with treatment based on a 13-item questionnaire. The overall score for each of five TSS domains (confidence to complete sexual activity, ease of erection, pleasure from sexual activity, erectile function satisfaction, and satisfaction with orgasm) was converted to a 0-100 scale with higher numbers on the scale indicating greater satisfaction. Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline TSS measurement, excluding those with International Index of Erectile Function - Erectile Function (IIEF-EF) domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 189 | 189 | 192
units on a scale
  Confidence to complete sexual activity | 27.0 (1.78) | 29.2 (1.78) | 3.8 (1.77)
  Ease of erection | 24.0 (1.69) | 24.7 (1.69) | 4.1 (1.68)
  Pleasure from sexual activity | 22.6 (1.58) | 22.7 (1.58) | 3.3 (1.57)
  Erectile function satisfaction | 31.0 (1.82) | 33.6 (1.81) | 4.9 (1.81)
  Satisfaction with orgasm | 25.6 (1.90) | 26.3 (1.89) | 6.2 (1.88)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for confidence to complete sexual activity. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 23.1, Standard Error of Mean 2.49
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 25.4, Standard Error of Mean 2.48
Statistical Analysis 3: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for ease of erection. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 19.9, Standard Error of Mean 2.36
Statistical Analysis 4: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 3]; LS Mean Difference = 20.6, Standard Error of Mean 2.35
Statistical Analysis 5: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for pleasure from sexual activity. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 19.3, Standard Error of Mean 2.21
Statistical Analysis 6: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 5]; LS Mean Difference = 19.5, Standard Error of Mean 2.20
Statistical Analysis 7: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for erectile function satisfaction. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 26.0, Standard Error of Mean 2.54
Statistical Analysis 8: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 7]; LS Mean Difference = 28.7, Standard Error of Mean 2.53
Statistical Analysis 9: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for satisfaction with orgasm. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 19.3, Standard Error of Mean 2.65
Statistical Analysis 10: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 9]; LS Mean Difference = 20.1, Standard Error of Mean 2.64

7. Secondary Outcome: Treatment Satisfaction Scale (TSS) - Patient Satisfaction With Medication Score at Week 12 Endpoint
Description: The TSS - patient satisfaction with medication measured participant satisfaction with treatment based on a 13-item questionnaire. The overall score was converted to a 0-100 scale with higher numbers on the scale indicating greater satisfaction. Satisfaction with medication was analyzed using analysis of covariance (ANOVA). The model included factors of study, treatment group, and pooled site within study.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline participant's satisfaction with medication measurement, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 189 | 189 | 192
units on a scale | 53.7 (1.98) | 55.9 (1.98) | 24.8 (1.97)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 28.9, Standard Error of Mean 2.77
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 31.0, Standard Error of Mean 2.76

8. Secondary Outcome: Change From Baseline to 12-Week Endpoint in the International Index of Erectile Function (IIEF) Question 15 (Sexual Confidence)
Description: Self-reported erectile function over the past 4 weeks. Question 15, confidence in the ability to get an erection, is scored from 1 (very low confidence) to 5 (very high confidence). Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline IIEF question 15 (Sexual Confidence) assessment, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 194 | 197 | 199
units on a scale | 1.2 (0.08) | 1.3 (0.08) | 0.3 (0.08)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 0.9, Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 1.0, Standard Error of Mean 0.11

9. Secondary Outcome: Change From Baseline to 12-Week Endpoint in Treatment Satisfaction Scale (TSS) - Partner
Description: The TSS measured participant's partner satisfaction with treatment based on a 13-item questionnaire. The overall score for each of five TSS domains (confidence to complete sexual activity, ease of erection, pleasure from sexual activity, erectile function satisfaction, and satisfaction with orgasm) was converted to a 0-100 scale with higher numbers on the scale indicating greater satisfaction. Least Squares (LS) mean of the change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model included centered-baseline as a covariate and factors of study, treatment group, and pooled site within study, and centered-baseline-by-treatment-group interaction.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline partner's TSS measurement, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 184 | 186 | 187
units on a scale
  Confidence to complete sexual activity | 23.7 (2.01) | 27.2 (1.99) | 2.0 (1.99)
  Ease of erection | 23.1 (1.76) | 25.3 (1.75) | 0.7 (1.75)
  Pleasure from sexual activity | 18.2 (1.69) | 18.5 (1.68) | 1.3 (1.68)
  Erectile function satisfaction | 28.6 (1.84) | 28.5 (1.83) | 3.4 (1.83)
  Satisfaction with orgasm | 18.7 (2.06) | 21.0 (2.05) | 3.6 (2.04)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 21.7, Standard Error of Mean 2.81
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; LS Mean Difference = 25.2, Standard Error of Mean 2.78
Statistical Analysis 3: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 3]; LS Mean Difference = 22.3, Standard Error of Mean 2.46
Statistical Analysis 4: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 3]; LS Mean Difference = 24.5, Standard Error of Mean 2.44
Statistical Analysis 5: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 5]; LS Mean Difference = 16.9, Standard Error of Mean 2.37
Statistical Analysis 6: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 5]; LS Mean Difference = 17.2, Standard Error of Mean 2.35
Statistical Analysis 7: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 7]; LS Mean Difference = 25.2, Standard Error of Mean 2.57
Statistical Analysis 8: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 7]; LS Mean Difference = 25.1, Standard Error of Mean 2.56
Statistical Analysis 9: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 9]; LS Mean Difference = 15.1, Standard Error of Mean 2.88
Statistical Analysis 10: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 9]; LS Mean Difference = 17.3, Standard Error of Mean 2.86

10. Secondary Outcome: Treatment Satisfaction Scale (TSS) - Partner Satisfaction With Medication Score at Week 12 Endpoint
Description: The TSS - partner satisfaction with medication measured participant's partner satisfaction with treatment based on a 13-item questionnaire. The overall score was converted to a 0-100 scale with higher numbers on the scale indicating greater satisfaction. Satisfaction with medication was analyzed using analysis of covariance (ANOVA). The model included factors of study, treatment group, and pooled site within study.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug, had a baseline and at least 1 post-baseline partner's satisfaction with medication measurement, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period III) | 5 mg Tadalafil (Period III) | Placebo (Period III)
Number analyzed (Participants) | 184 | 186 | 187
units on a scale | 52.5 (1.97) | 55.7 (1.96) | 27.5 (1.96)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 25.1, Standard Error of Mean 2.76
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period III) vs Placebo (Period III); Test type: Superiority or Other; p < 0.001, ANOVA — Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted; LS Mean Difference = 28.2, Standard Error of Mean 2.74

11. Secondary Outcome: Percentage of Participants Having International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score Greater Than or Equal to 26 From 12 to 16 Weeks
Description: Self-reported erectile function over the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Data presented are the percentage of participants who return to normal erectile function (IIEF-EF domain score ≥26) at end of open-label extension treatment period (Period IV).
Time Frame: 12 weeks through 16 weeks
Population: All participants who were entered the open-label treatment, received at least 1 dose of study drug during open-label treatment, had Week 12 and at least 1 IIEF-EF measurement during open-label treatment, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Number; unit: percentage of participants
Groups:
- 2.5 mg Titrated to 5 mg Tadalafil (Period IV): 5.0 milligram (mg) Tadalafil for 4 weeks during open-label extension treatment period (Period IV).
- 5 mg Tadalafil (Period IV); Placebo (Period IV): 5.0 mg Tadalafil for 4 weeks during open-label extension treatment period (Period IV).
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period IV) | 5 mg Tadalafil (Period IV) | Placebo (Period IV)
Number analyzed (Participants) | 178 | 179 | 183
percentage of participants | 54.5 | 59.8 | 62.8

12. Secondary Outcome: Change From 12 Weeks to 16 Weeks in Participant's International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score
Description: Self-reported erectile function over the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function.
Time Frame: 12 weeks and 16 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period IV) | 5 mg Tadalafil (Period IV) | Placebo (Period IV)
Number analyzed (Participants) | 178 | 179 | 183
units on a scale
  End of Week 12 | 22.4 (6.71) | 22.5 (7.07) | 16.0 (7.39)
  End of Week 16 | 24.1 (6.44) | 24.2 (6.46) | 24.4 (6.73)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period IV); Test type: Superiority or Other; p < 0.001, Paired t-test — Comparison of Week 16 to Week 12. Sequential gatekeeping strategies were applied for multiplicity control and the p-value was not adjusted
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period IV); Test type: Superiority or Other; p < 0.001, Paired t-test — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Placebo (Period IV); Test type: Superiority or Other; p < 0.001, Paired t-test — [p-value comment as in outcome 12, analysis 1]

13. Secondary Outcome: Change From Week 12 to Week 16 Percentage of "Yes" Responses to Sexual Encounter Profile (SEP) Questions 3
Description: Assessed the percentage of Yes responses to the SEP diary Question 3 "Did your erection last long enough for you to have successful intercourse?" from Week 12 (end of double-Blind treatment) to Week 16 (end of open-label treatment).
Time Frame: 12 weeks and 16 weeks
Population: All participants who were entered the open-label treatment, received at least 1 dose of study drug during open-label treatment, had Week 12 and at least 1 SEP diary Question 3 measurement during open-label treatment, excluding those with IIEF-EF domain score ≥26 ("normal") at baseline. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: percentage of "yes" responses
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil (Period IV) | 5 mg Tadalafil (Period IV) | Placebo (Period IV)
Number analyzed (Participants) | 176 | 177 | 181
percentage of "yes" responses
  End of Week 12 | 68.3 (38.25) | 69.0 (37.88) | 43.1 (39.03)
  End of Week 16 | 75.0 (34.49) | 75.5 (34.89) | 80.0 (34.37)
Statistical Analysis 1: Comparison: 2.5 mg Titrated to 5 mg Tadalafil (Period IV); Test type: Superiority or Other; p = 0.002, Paired t-test — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: 5 mg Tadalafil (Period IV); Test type: Superiority or Other; p = 0.004, Paired t-test — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Placebo (Period IV); Test type: Superiority or Other; p < 0.001, Paired t-test — [p-value comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Arm/Group | 2.5 mg Titrated to 5 mg Tadalafil | 5 mg Tadalafil | Placebo | 5 mg Tadalafil Open-Label Extension
Serious Adverse Events (participants affected / at risk) | 1/205 | 1/205 | 1/207 | 3/546
Other Adverse Events (participants affected / at risk) | 46/205 | 68/205 | 50/207 | 23/546
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg Titrated to 5 mg Tadalafil (N=205) | 5 mg Tadalafil (N=205) | Placebo (N=207) | 5 mg Tadalafil Open-Label Extension (N=546)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg Titrated to 5 mg Tadalafil (N=205) | 5 mg Tadalafil (N=205) | Placebo (N=207) | 5 mg Tadalafil Open-Label Extension (N=546)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure via father (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytology abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 1 (1) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 4 (4) | 9 (9) | 7 (8) | 4 (4)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organic erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia of genital male (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dental care (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days